CLINICAL TRIAL: NCT05137964
Title: Is Vitamin D The Missing Piece of the Subfertility Puzzle in Pakistani Women? A Cross Sectional Evaluation of Vitamin D Status and Ovarian Reserve Markers
Brief Title: A Cross Sectional Evaluation of Vitamin D Status and Ovarian Reserve Markers
Status: Completed | Type: Observational
Sponsor: Australian Concept Medical Center (Other)
Responsible Party: Principal Investigator, Uzma Imran, Consultant Gyn Obs, Australian Concept Medical Center
Other Study IDs: 2021-07-01-Uzma Imran
Record Dates: First submitted 2021-11-05; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Subfertility, Female
Keywords: subfertile; female
MeSH Terms: conditions — Infertility, Female | interventions — Vitamin D Response Element

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin D Deficient: deficiency (<20ng/ml)
  Interventions: Diagnostic Test: Vitamin D
- Vitamin D Sufficient: sufficiency (>30ng/ml)
  Interventions: Diagnostic Test: Vitamin D

INTERVENTIONS:
Diagnostic Test: Vitamin D — Serum Biochemical routine lab workup and gynaecological ultra sound AFC
  Other Names: Serum AMH, 25-hydroxyvitamin D (25-OHD), FSH and Antral Follicle Count (AFC) via ultra sound

SUMMARY:
Evaluation of the association between vitamin D (VD) deficiency and ovarian reserve markers in a group of Pakistani sub fertile women was conducted

DETAILED DESCRIPTION:
Objective

This study was conceived with the objective to assess ovarian reserves in presence of vitamin D deficiency (VDD) in a select group of Pakistani sub fertile women, presenting at a specialized fertility centre. The measurements of antral follicle count (AFC), Serum Anti-Müllerian hormone (AMH), Serum Follicle-stimulating hormone (FSH) and Serum Vitamin D (VD) levels were the main tools used for the assessment of ovarian reserve.

Materials & Methods A retrospective cross-sectional study was conducted at the Australian Concept Medical Centre after approval from the institutional ethical review committee. All female patients aged 18 to 45 years, presenting with primary and/or secondary subfertility, at the Australian Concept Medical Centre in Karachi, Pakistan from August 2016 to July 2021 were included in the study (n=301). Inclusion criteria was focused on subjects labelled as sub fertile by the consultant gynecologist, based on the criteria of failed to conceive after 12 months of no contraceptive use. Patients with missing data i.e., BMI, duration of subfertility, age, AMH, 25-hydroxyvitamin D (25-OHD), AFC and FSH were further excluded.

The Biochemical analysis was performed at the section of Chemical Pathology, department of Pathology and Laboratory Medicine, Aga Khan University, Karachi. 25-OHD was analyzed by a chemiluminescence assay on the liaison XL (DiaSorin) analyzer. AMH was measured using electro chemiluminescence assay on the Roche Diagnostic e411 analyzer. While FSH quantification was done using ADVIA Centaur FSH assay from Siemens Medical Solutions Diagnostics USA. The internal and external quality assurance was ensured according to the institutional protocol. Moreover, the laboratory is accredited by the College of American Pathologists (CAP) and Joint Commission international, ensuring external quality assurance.

AFC was determined through a transvaginal 2D ultrasound of the pelvis. To reduce the bias, all ultrasound scans were conducted in the center using the same machine (Model 6v1: Sonoscape) and vaginal probe (3.5 Hz). Before ultra sound procedure, patients were directed to empty bladder and a standard ultrasound technique was used. Two values were obtained, one for each ovary, and an average was taken to obtain a final value.

The data of all eligible patients was recorded in the pre-defined Performa designed for this study. The Kruskal-Wallis Test and one way ANOVA was applied to report the distribution of the data. The correlation between the categorical variables (25-OHD levels with AFC and AMH) was assessed using the Chi-Square test and Spearman Correlation. Comparison was based on 25-OHD levels grouped into three categories: deficiency (<20ng/ml), insufficiency (21-29 ng/ml) and sufficiency (>30ng/ml). AMH was categorized as low (<1 ng/ml), low normal (1-2 ng/ml), normal (2-4 ng/ml), and high (>4 ng/ml). The third variable, AFC, was also classified into very low (<6), low normal (6-8), normal (8-10), high normal (10-12), very high (>12). The p value <0.05 was considered statistically significant. The statistical analysis was performed using the statistical software IBM SPSS Statistics for Windows version 23.0 (IBM Corp. Released 2015. Armonk, NY: IBM Corp).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary and/or secondary subfertility

Exclusion Criteria:

* Patients with missing data i.e., BMI, duration of subfertility, age, AMH, 25-hydroxyvitamin D (25-OHD), AFC and FSH.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pakistani female patients aged 18 to 45 years, presenting with primary and/or secondary subfertility
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation | Aug 2016 to July 2021
  To address gaps in local data, this study was conducted to explore the association between VDD and ovarian reserve, via measurements of AFC, AMH, FSH and 25-hydroxy vitamin D (25-OHD) in Pakistani women.

IPD SHARING:
Plan to Share IPD: No